CLINICAL TRIAL: NCT04473326
Title: Optimizing Message Framing for Healthy Habits for Patients With Type 2 Diabetes - Phase II (Pragmatic Trial)
Brief Title: Reinforcement Learning in Diabetes Mellitus Trial
Acronym: REINFORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julie Lauffenburger, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020P000846; P30AG064199-01 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence | interventions — Reinforcement Machine Learning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforcement Learning Intervention Arm (Experimental): Up to daily, tailored text messages.
  Interventions: Behavioral: Reinforcement Learning
- Control Arm (No Intervention): Up to daily, untailored text messages.

INTERVENTIONS:
Behavioral: Reinforcement Learning — Participants in the intervention arm will receive up to daily, tailored text messages based on their electronic pill bottle-measured adherence. Given the participants' baseline characteristics and time-varying responses to the messages, a reinforcement learning algorithm will deliver different text messages and adapt over time to determine which type of messaging works best for each individual participant.
  Arms: Reinforcement Learning Intervention Arm

SUMMARY:
Reinforcement learning is an advanced analytic method that discovers each individual's pattern of responsiveness by observing their actions and then implements a personalized strategy to optimize individuals' behaviors using trial and error. The goal of this pilot study is to develop and test a novel reinforcement learning-enhanced text messaging program to support medication adherence in patients with type 2 diabetes. Type 2 diabetes is an optimal condition in which to test this program, as it is one of the most prevalent chronic conditions in the US adult population and requires most patients to be on daily or twice daily doses of medications. This pilot study will be a parallel randomized pragmatic trial comparing medication adherence and clinical outcomes for adults aged 18-84 with type 2 diabetes who are prescribed 1-3 daily oral medications for this disease. Participants will be randomized to one of two arms for the duration of the study period: (1) a reinforcement learning intervention arm with up to daily, tailored text messages based on time-varying treatment-response patterns; or (2) a control arm with up to daily, un-tailored text messages. Our outcomes of interest will be medication adherence, as measured by electronic pill bottles, and HbA1c levels.

DETAILED DESCRIPTION:
The goal of this pilot study is to develop and test a novel reinforcement learning-enhanced text messaging program to support medication adherence in patients with type 2 diabetes. This pilot study will be a parallel randomized pragmatic trial comparing medication adherence and clinical outcomes for adults aged 18-84 with type 2 diabetes who are prescribed 1-3 daily oral medications for this disease. Participants will be randomized to one of two arms for the duration of the study period: 1) a reinforcement learning intervention arm with up to daily, tailored text messages based on time-varying treatment response patterns, or 2) a control arm with up to daily, untailored text messages. Our outcomes of interest will be medication adherence, as measured by electronic pill bottles, and HbA1c levels.

ELIGIBILITY:
Inclusion criteria:

* Age between 18-84 years
* Diagnosed with type 2 diabetes mellitus (T2DM) and are prescribed between 1-3 daily oral medications for this disease
* Currently have a smartphone with a data plan or WiFi at home
* HbA1c level ≥7.5%
* Basic working knowledge of English
* Willing and able to set up the platform and adhere to study procedures
* Either not currently using a pillbox or willing to use electronic pill bottles (EDMs) for diabetes medications for the duration of the study

Exclusion criteria:

* Patients with active enrollment in another diabetes trial within Mass General Brigham
* Patients who receive daily assistance with taking their medications at home
* Patients who are unable to receive text messages for more than 3 days in a row during the study period

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lauffenburger JC, Yom-Tov E, Keller PA, McDonnell ME, Bessette LG, Fontanet CP, Sears ES, Kim E, Hanken K, Buckley JJ, Barlev RA, Haff N, Choudhry NK. REinforcement learning to improve non-adherence for diabetes treatments by Optimising Response and Customising Engagement (REINFORCE): study protocol of a pragmatic randomised trial. BMJ Open. 2021 Dec 3;11(12):e052091. doi: 10.1136/bmjopen-2021-052091. PMID 34862289

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reinforcement Learning Intervention Arm | Control Arm
Started | 29 | 31
Completed | 28 | 28
Not Completed | 1 | 3
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reinforcement Learning Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.31 (11.35) | 56.68 (12.89) | 58.43 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 17 | 17 | 34
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Self-reported automaticity of medication-taking, n(%) [Count of Participants; unit: Participants] — Higher scores are better (i.e., higher automaticity indicates that respondents think that medication-taking is more automatic) based on a self-reported measure of automaticity
  Participants
    0-1 (no or low automaticity) | 7 | 12 | 19
    2+ (high automaticity) | 22 | 19 | 41
Baseline HbA1c, mean (sd) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.99 (1.39) | 9.10 (1.47) | 9.05 (1.42)
Education level, n(%) [Count of Participants; unit: Participants]
  High school graduate or below | 7 | 5 | 12
  Some college/college graduate | 15 | 19 | 34
  Post-graduate | 7 | 7 | 14
Number of self-reported physicians, n(%) [Count of Participants; unit: Participants]
  1-3 | 10 | 15 | 25
  4+ | 19 | 16 | 35
Number of self-reported medications, n(%) [Count of Participants; unit: Participants]
  1 | 2 | 2 | 4
  2-4 | 6 | 4 | 10
  5+ | 21 | 25 | 46
Number of Pillsy bottles, n(%) [Count of Participants; unit: Participants]
  1 | 20 | 25 | 45
  2+ | 9 | 6 | 15
Level of non-adherence, self-reported number of doses missed in past month, n(%) [Count of Participants; unit: Participants]
  0 | 12 | 14 | 26
  1+ | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Medication adherence to type 2 diabetes oral medications (averaged) as measured by the number of dates and times of pillbottle openings in the electronic pill bottles
Time Frame: 6 months
Population: Participants were included in the analysis until they no longer participated in the study.
Measure: Mean (Standard Deviation); unit: pill bottle openings
Arm/Group | Reinforcement Learning Intervention Arm | Control Arm
Number analyzed (Participants) | 29 | 31
pill bottle openings | 74 (31) | 68 (29)

2. Secondary Outcome: Glycemic Control
Description: Change in glycated hemoglobin A1c from baseline to end of the 6-month follow-up
Time Frame: 6 months
Population: Participants were included in the analysis until they no longer participated in the study. Differences were calculated among those who had follow-up HbA1c values recorded.
Measure: Mean (Standard Deviation); unit: percentage glycated hemoglobin
Arm/Group | Reinforcement Learning Intervention Arm | Control Arm
Number analyzed (Participants) | 29 | 31
percentage glycated hemoglobin | -0.82 (1.19) | -1.20 (2.28)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through the 6 month study follow-up period.
Arm/Group | Reinforcement Learning Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04473326/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT04473326/ICF_000.pdf